CLINICAL TRIAL: NCT01823588
Title: Efficacy of a Nurse-led Reminder Program for the Management of the Risk Factors for Cardiovascular Diseases in Hypertensive Patients: a Randomized Controlled Trial
Brief Title: Nurse-led Reminder Program for the Prevention of Cardiovascular Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi 'G. d'Annunzio' Chieti e Pescara (Other)
Responsible Party: Principal Investigator, Lamberto Manzoli, Associate Professor of Epidemiology and Public Health, Università degli Studi 'G. d'Annunzio' Chieti e Pescara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Nurse led
Record Dates: First submitted 2013-03-28; First posted 2013-04-04 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Hypertension; Cardiovascular Disease
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention): Educational program and usual cardiovascular prevention.
- Nurse-led reminder through email (Experimental): In addition to usual care and educational program, the intervention group will also receive email alerts and phone calls from the nurse-care manager (NCM)
  Interventions: Behavioral: Nurse-led reminder through email.

INTERVENTIONS:
Behavioral: Nurse-led reminder through email. — Both groups will receive an educational program and usual care. The educational program will consist of 1-hour sessions, during which the NCM emphasize the importance of blood pressure control and correct measurement, give advice for a correct blood pressure self-measurement; report non-pharmacological strategies for a healthy lifestyle, and instruction on how to fill the daily self-assessment form.
  Educational program and usual cardiovascular prevention. The educational program will consist of 1-hour sessions, during which the NCM emphasize the importance of blood pressure control and correct measurement, give advice for a correct blood pressure self-measurement; report non-pharmacological strategies for a healthy lifestyle, and instruction on how to fill the daily self-assessment form.
  Arms: Nurse-led reminder through email

SUMMARY:
A number of strategies have been evaluated to improve the prevention and control of the main cardiovascular (CVD) risk factors. Nursing telephonic and tele-counseling individualized lifestyle educational programs were found to improve blood pressure (BP) control and adherence to healthy lifestyle. This study aims at evaluating for the first time the efficacy of a nurse-led reminder program through email (NRP-e) to improve CVD risk factors among hypertensive adults.

Participants will receive usual care and a guideline-based educational program on BP control and healthy lifestyle habits. Subjects in the NRP-e group will also receive weekly email alerts and phone calls from a nurse care manager for 6 months. Emails contain a reminder program on the compliance with a healthy lifestyle based upon current guidelines for CVD prevention. Follow-up visits will be scheduled at 1, 3 and 6 months after enrollment; randomization will be made centrally and blood samples will be evaluated into a single, accredited laboratory.

ELIGIBILITY:
Inclusion Criteria:

* to be eligible, all subjects had to be hypertensive (on active treatment for hypertension, or systolic blood pressure ≥ 140 mmHg; or
* diastolic blood pressure ≥ 90 mmHg).
* speaking and reading Italian,
* having a active phone number and an email address, and
* providing a signed informed consent.

Exclusion Criteria:

* mental illness;
* nursing home institutionalization;
* pregnancy;
* previous cardiovascular major events, non-modifiable cardiovascular risk-factors (i.e. diabetes).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2013-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The main outcome of the study was the mean difference between groups in the average reduction in systolic and diastolic blood pressure between baseline and the end of follow-up | 6 months

SECONDARY OUTCOMES:
Mean difference between groups in the average reduction in LDL cholesterol between baseline and the end of follow-up | 6 months
Mean difference between groups in the average reduction in physical activity between baseline and the end of follow-up | 6 months
Mean difference between groups in the average reduction in BMI between baseline and the end of follow-up | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo GC Cicolini, PhD, Principal Investigator — ASL 02 Abruzzo - Abruzzo Region - Italy
Locations (2):
- Italy (2):
  - ASL02Abruzzo, Chieti, Abruzzo
  - Department of Medicine and Aging Sciences, University of Chieti, Chieti, CH

REFERENCES:
- [Result] Cicolini G, Simonetti V, Comparcini D, Celiberti I, Di Nicola M, Capasso LM, Flacco ME, Bucci M, Mezzetti A, Manzoli L. Efficacy of a nurse-led email reminder program for cardiovascular prevention risk reduction in hypertensive patients: a randomized controlled trial. Int J Nurs Stud. 2014 Jun;51(6):833-43. doi: 10.1016/j.ijnurstu.2013.10.010. Epub 2013 Oct 25. PMID 24225325